CLINICAL TRIAL: NCT02429297
Title: Developing Accessible Telehealth Programs for Diabetes and Hypertension Management in Bolivia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, VA Senior Research Career Scientist, Professor of Health Behavior and Health Education and of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00081734
Record Dates: First submitted 2015-03-04; First posted 2015-04-29 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension; Diabetes
Keywords: Hypertension; Diabetes; mHealth; Interactive Voice Response; Bolivia; Chronic disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patient Only - HITCM-only (Experimental): Patients enrolling without a CarePartner receive weekly Health Information Technology/Care Manager (HITCM) automated assessment and self-care support calls with feedback to the clinical team.
  Interventions: Other: HITCM-only
- Patient & CarePartner - HITCM-only (Experimental): Patients enrolling with a CarePartner receive weekly Health Information Technology/Care Manager (HITCM) automated assessment and self-care support calls with feedback to the clinical team.
  Interventions: Other: HITCM-only
- Patient & CarePartner - HITCM+CP (Experimental): Patients enrolling with a CarePartner receive weekly Health Information Technology/Care Manager (HITCM) automated assessment and self-care support calls with feedback to the clinical team plus updates to their CarePartner via phone or email.
  Interventions: Other: HITCM+CP

INTERVENTIONS:
Other: HITCM-only — HITCM-only group: patients receive weekly automated calls with feedback to the clinical team.
  Arms: Patient & CarePartner - HITCM-only; Patient Only - HITCM-only
Other: HITCM+CP — HITCM + CP group: patients receive weekly automated calls with feedback to the clinical team and their CarePartner receives updates via phone or email.
  Arms: Patient & CarePartner - HITCM+CP

SUMMARY:
The purpose of the study is to evaluate the feasibility and impact of an automated phone system in monitoring and improving self-care and health outcomes among patients with diabetes and/or hypertension in Bolivia, in addition to assessing the additional benefit of support from a family member or friend.

DETAILED DESCRIPTION:
All patients will receive weekly automated calls with feedback to the clinical team. Blood pressures will be taken for all patients by researchers and finger-stick blood glucose readings will be taken at baseline for diabetic patients only and if possible, at follow-up. Fingersticks will use the patient's own glucometer or standard home glucometers donated by the project to the clinic. Patients will be informed about their blood pressure results; and, the clinic will be alerted if the systolic BP exceeds 150.

If participants enroll with a CarePartner, they will be randomized to have their CarePartner receive weekly automated updates focused on symptom monitoring and patient self-care (HITCM+CP) versus usual care (no updates to CarePartner), HITCM-only. All participants will receive a weekly 10-15 minute automated phone call to their cell phone for disease assessment and self-care support for up to 16 weeks. Some patients with hypertension may be provided with in-home cuffs for measurement of blood pressure throughout the study. During enrollment, the research team will explain how the cuffs are used, as well as how to work the automated phone system. During patients' automated calls, they will be asked questions about their self-care relevant to their diagnosis, blood pressure regimen and readings (hypertension only), diet, glucose monitoring and symptoms of high/low blood sugar (diabetes only) and medication adherence. Based on the patient's self-report, they will receive targeted suggestions for how to improve their self-management. No identifying information is included in the automated call sent to the patient's phone other than the patient's first name. At the end of each automated call, patients will hear the phone number of their clinic, which they can call for a health problem or to disenroll from the program. At the time of recruitment, an initial automated call will be sent to the patient's phone so that they can learn what to expect and have the chance to ask questions of the research associate.

In the event that the patient reports a health or self-care problem during their call (i.e., the patient reports rarely or never taking their medication), a report will automatically be generated and sent by email to the research team plus the patient's designated clinician so that follow-up can take place. The secure email address will be verified with each clinician, and be password protected.

The intervention will last up to 16 weeks, after which the patient will have a follow-up meeting with the research team and will complete a survey about the program. All follow-ups will take place either in person or over the phone. Patients will receive an incentive at follow-up at no more than $10 USD.

ELIGIBILITY:
Inclusion Criteria:

* 21-80 years of age
* Diagnosis of hypertension, a systolic blood pressure > 140mmHg, and/or diagnosis of diabetes
* Access to a functional cell phone
* Able to respond to automated telephone calls

Exclusion Criteria:

* Life-threatening health problem such as cancer with less than a six month life expectancy
* Are visiting the clinic for an urgent health problem (for themselves)
* If they have severe mental illness as reported by their clinical team

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline on self-care behaviors and health at 16 weeks (questionnaire) | Up to 16 weeks

SECONDARY OUTCOMES:
Patient satisfaction (satisfaction questionnaire) | Up to 16 weeks
Evaluate program feasibility (questionnaire, satisfaction, and usage rates) | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (1):
- El Servicio Departmental de Salud (SEDES) affiliated clinics, La Paz, Bolivia

IPD SHARING:
Plan to Share IPD: No